CLINICAL TRIAL: NCT05491317
Title: A Phase 1 Dose Finding and Phase 2, Randomized, Open-Label Trial to Evaluate the Safety and Clinical Activity of Immunoradiotherapy Combinations as a Treatment Option in Subjects With Metastatic Solid Tumors
Brief Title: A Safety and Antitumor Activity Trial of Immunoradiotherapy Combinations as a Treatment Option for Subjects With Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: After reviewing all available data from Part 1 of the trial, the Sponsor has decided not to proceed to Part 2 (randomized Phase 2) of the trial due to lack of efficacy
Sponsor: Genmab (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1042-02; 2022-000509-29 (EudraCT Number); 2023-508529-29-00 (EU CTIS Number); RECF-005058 (Registry Identifier: National Institute of Cancer France)
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Non-CNS Tumor
MeSH Terms: interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Part 1 is sequential, Part 2 is parallel (randomized)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Radiotherapy + GEN1042 (Experimental)
  Interventions: Biological: GEN1042; Radiation: Radiotherapy
- Radiotherapy + GEN1042 + Pembrolizumab (Experimental)
  Interventions: Biological: GEN1042; Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Biological: GEN1042 — Intravenous
Drug: Pembrolizumab — Intravenous
  Arms: Radiotherapy + GEN1042 + Pembrolizumab
Radiation: Radiotherapy — Radiotherapy

SUMMARY:
The main purpose is to assess the safety and clinical activity of GEN1042 in combination with radiotherapy or GEN1042 in combination with radiotherapy and pembrolizumab as a treatment option for participants with metastatic solid tumors.

DETAILED DESCRIPTION:
The study will be conducted in two parts: Part 1 (dose-finding) and Part 2 (randomization).

Part 1 will evaluate the safety of immunoradiotherapy combinations and establish the dose(s) to be evaluated in Part 2.

Part 2 will evaluate the anti-tumor activity of immunoradiotherapy combinations at the established dose(s) from Part 1.

Participants in both parts are treated with one of the following combinations:

* Radiotherapy + GEN1042
* Radiotherapy + GEN1042 + Pembrolizumab

While participants in Part 1 are assigned sequentially (GEN1042 without pembrolizumab is investigated first), participants in Part 2 are randomized 1:1 in the two treatment arms.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with histologically confirmed non-central nervous system (CNS) solid tumor that is metastatic and for whom there is no available standard therapy.
* At least 18 years of age.
* Signed informed consent prior to any screening procedures.
* Measurable disease according to RECIST v1.1.
* Life expectancy of >3 months.
* Qualify for palliative radiotherapy as an available option for disease management.
* Eastern Cooperative Oncology Group (ECOG) 0-1.
* Normal or adequate liver, renal, cardiac and bone marrow function.

Key Exclusion Criteria:

* Prior malignancy except for non-melanoma skin cancers and in situ cancers.
* Condition contraindicating radiotherapy.
* Rapidly progressing disease.
* Active, known or suspected autoimmune disease.
* History of non-infectious pneumonitis that required steroids or currently has pneumonitis.
* Contraindications to the use of pembrolizumab.
* Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of first treatment.
* Received an allogeneic tissue/solid organ transplant.
* Active infection requiring systemic therapy.

Note: Other protocol defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose Limiting Toxicities (DLTs) | During the first cycle (Cycle length = 21 days)
  Toxicities will be graded for severity according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0).
Part 2: Number of Participants with Abscopal Response in Non-irradiated Target Lesions | Up to 12 months after the last radiation treatment
  Assessed by investigator.

SECONDARY OUTCOMES:
Parts 1 and 2: Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST) v1.1 as assessed by investigator.
Parts 1 and 2: Duration of Response (DOR) | Up to 2 years
  DOR is defined as the time from the onset date of response to the date of the first documented progression or death due to any cause based on RECIST v1.1 as assessed by investigator.
Parts 1 and 2: Disease Control Rate (DCR) | Up to 2 years
  The disease control rate (DCR) is defined as the percentage of participants with BOR of CR, PR, and stable disease (SD) according to RECIST v1.1.
Parts 1 and 2: Progression Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the date of randomization (or date of first administration of GEN1042 ± pembrolizumab treatment for participants in Part 1) to the date of the first documented progression or death due to any cause based on RECIST v1.1 as assessed by investigator.
Parts 1 and 2: One- year Overall Survival (OS) | Up to 2 years
  OS is defined as the time from date of randomization (or date of first administration of GEN1042 ± pembrolizumab treatment for participants in Part 1) to date of death due to any cause.
Part 1: Number of Participants With Abscopal Response in Non-irradiated Target Lesions | Up to 12 months after the last radiation treatment
  Assessed by investigator.
Parts 1 and 2: Number of Participants with Adverse Events (AEs) | From screening until the end of the safety follow-up period (30 days or 90 days after last dose)
Parts 1 and 2: Area Under the Concentration-time Curve (AUC) of GEN1042 | Predose and postdose at multiple timepoints up to 30 days after last dose
Parts 1 and 2: Maximum (Peak) Plasma Concentration (Cmax) | Predose and postdose at multiple timepoints up to 30 days after last dose
Parts 1 and 2: Elimination Half-life (T1/2) of GEN1042 | Predose and postdose at multiple timepoints up to 30 days after last dose
Parts 1 and 2: Number of Participants with Anti-drug Antibodies (ADAs) | Predose at multiple timepoints up to 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (3):
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No